CLINICAL TRIAL: NCT02981654
Title: Prospective, Open-Label, Multi-Center, Non- Comparative Study to Assess the Safety and Efficacy of CO2 Laser System (FemiLiftTM) in the Treatment of Stress Urinary Incontinence (SUI) in Female Subjects.
Brief Title: Safety and Efficacy of Carbone Dioxide (CO2) Laser System in Treatment of Female Stress Urinary Incontinence.
Acronym: CO2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Collaborators: The Baruch Padeh Medical Center, Poriya (Other Government); Kaplan Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2092-15-SMC
Record Dates: First submitted 2016-10-30; First posted 2016-12-05 (Estimated); Last update posted 2016-12-06 (Estimated); Status verified 2016-12

CONDITIONS: Female Stress Urinary Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Femilift treatment (Experimental): The Alma Lasers Pixel carbon dioxide laser system delivers fractionated laser energy through a special lens that divides the energy into a 9 x 9 (81) matrix of 1 cm square area. The fractional laser rays cause thermal damage that reaches the vaginal sub - epithelium to stimulate the growth of new collagen.
  Intervention: FemiLift vaginal handpiece is inserted into the vagina, to deliver CO2 laser energy. The vaginal epithelium is covered by rotation of vaginal handpiece in 360 degrees, releasing laser energy at 6-8 points, and than withdrawn 1 cm each time to perform the same process, to cover the the total vaginal length.
  Interventions: Device: Alma Lasers Pixel carbon dioxide laser system

INTERVENTIONS:
Device: Alma Lasers Pixel carbon dioxide laser system — The vaginal handpiece sheath is lubricated with baby oil. Set the initial energy level (startup set up recommendations: High mode, 40 millijoule/pixel; according to the patient reaction you can increase up to 120 max. Pulse mode or Repeat mode). The handpiece is inserted as distally as possible, with the laser energy's window oriented to the 12:00 o'clock position. There are position markings on the handpiece. Trigger a laser pulse by pressing the footswitch. Shoot the laser and rotate the probe by one hour at a time. When you reach the 12:00 o'clock position again, withdrawal the headpiece back by one centimeter and repeat the rotational treatment process.

SUMMARY:
This is a prospective, open-label, multi-center, non-comparative study that will be conducted on female subjects between 30 and 75 years of age, diagnosed with stress urinary incontinence (SUI).

Following the screening period, including urodynamic assessment to confirm SUI, each subject will undergo three FemiLiftTM treatment sessions, and will be followed up for a period of one year. The main efficacy endpoint in this study is defined as significant improvement (score of 6 or 7) in the urinary incontinence measured with PGI-I score at the 6 months visit. Various subjective and objective measures of incontinence severity, quality of life, sexual function and tissue effects will be performed at follow up.

DETAILED DESCRIPTION:
Improvement in SUI symptoms as measured by the following parameters:

Objective parameters:

* Change from baseline in 3 days Urinary Diary - at 1, 2, 6 and 12 months:

  * Number of incontinence episodes per day
  * Number of pads used per day
* Change from baseline in 1 hour pad test 1, 2, 6 and 12 months
* Change from baseline as assessed with Vaginal Biopsy

Subjective parameters:

* Patient Global Impression of Severity (PGI-S) - 4-point Likert scale - at screening, 1, 2, 6 and 12 months
* Change from baseline in Pelvic Floor Distress Inventory Questionnaire (PFDI) - at 1, 2, 6 and 12 months
* Change from baseline in Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire (PISQ) - at 1, 2, 6 and 12 months
* Change from baseline in Pelvic Floor Impact Questionnaire (PFIQ) - at 1, 2, 6 and 12 months

ELIGIBILITY:
Inclusion Criteria:

* Females between 30 and 75 years of age
* Provided written Informed Consent
* Patients with mild to moderate stress urinary incontinence (SUI) [according to the severity index developed by Sandvik]
* Patients with mixed urinary incontinence, while the predominant symptoms are stress related, may also be enrolled
* Normal Papanicolaou smear (up to 1 year prior to screening)
* Negative urine culture
* Vaginal canal, introitus and vestibule free of injuries and bleeding
* Positive urinary stress test (Urine leakage is demonstrated while the patient is examined with full bladder in lithotomy position, and asked to perform 3 strong coughs).

Exclusion Criteria:

* Positive pregnancy test
* Planned pregnancy within the next year
* Severe prolapse (POP>= grade 3)
* Use of photosensitive drugs
* Injury or/and active infection in the treatment area
* Active vaginal infection
* human papillomavirus/herpes simplex virus
* Undiagnosed vaginal bleeding
* Urge or overflow incontinence
* Patients who are on antidepressants, or α-adrenergic and anticholinergic medications
* Patients with immune system diseases.
* Patients with allergic reaction to laser.
* Patient under treatment with photosensitivity side effects medication.
* Obese women (BMI >30)
* Patient unable to follow post treatment instructions.

Ages: 30 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-12; Primary Completion 2017-05 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Success Rate - SUI Symptom Improvement | 6 months
  Success rate - defined as an improvement in SUI symptoms as a score or 6 or 7 measured by the Patient Global Impression of Improvement (PGI-I) - 7-point Likert scale - at the 6 months visit

SECONDARY OUTCOMES:
Urinary Diary | 12 months
  Change from baseline in 3 days Urinary Diary - at 1, 2, 6 and 12 months post first treatment:
  * Number of incontinence episodes per day
1 hour pad test | 12 months
  Change from baseline in 1 hour pad test at 1, 2, 6 and 12 months post first treatment
Vaginal Biopsy | 12 months
  Sample will be obtained from the vaginal mucosa 2 cm inside the introitus on the lateral vaginal wall.
PGI-S | 12 months
  Change from baseline in Patient Global Impression of Severity (PGI-S) over time
PFDI | 12 months
  Change from baseline in Pelvic Floor Distress Inventory Questionnaire (PFDI) over time
PISQ | 12 months
  Change from baseline in Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire (PISQ) over time
PFIQ | 12 months
  Change from baseline in Pelvic Floor Impact Questionnaire (PFIQ) over time
Safety Endpoint assessed by the rate of serious device related adverse events | 12 months
  The rate of serious device related adverse events reported during the study

CONTACTS AND LOCATIONS:
Overall Officials: Menachem Alcalay, MD, Principal Investigator — Head, Urogynecology Unit, Chaim Sheba Medical Center

IPD SHARING:
Plan to Share IPD: No